CLINICAL TRIAL: NCT01237158
Title: Genetic Association Study Between GAD1 and Reelin Polymorphisms and GABA/Glutamate MRS in Bipolar Disorder Type 1 and Healthy Controls: SPECGENE PROJECT
Acronym: SPECGENE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Ricardo Alberto Moreno, University of Sao Paulo
Other Study IDs: nov 2010
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2010-10

CONDITIONS: Bipolar Disorder
Keywords: GAD1,; GAD67,; bipolar,; GABA,; Glutamate,; Reelin,; Rln,; Spectroscopy; euthymic bipolar I patients
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- healthy controls
- bipolar disorder type I

SUMMARY:
Background: The pathophysiological mechanisms of bipolar disorder are not completely clarified and several hypothesis have already been formulated including the role of monoamines, gama amino butyric acid (GABA) and glutamate. GABA is the main inhibitory neurotransmitter while glutamate is the main excitatory neurotransmitter. Genes that play a role in GABA metabolism and in the activity of GABA neurons are very important to understand the GABA function, once they affect neurodevelopment and its dysfunctions may predispose to neuropsychiatric diseases. The two genes that are going to be study in this project are glutamic acid decarboxylase (GAD1) and reelin (Reln). The enzyme glutamic acid descarboxylase (GAD67) metabolizes glutamate in GABA in the pre synaptic neuronal regions and is coded by the gene GAD1. Reelin is secretory serine protease with dual roles in mammalian brain: embryologically, it guides neurons and radial glial cells to their corrected positions in the developing brain; in adult brain, Reelin is involved in a signaling pathway which underlies neurotransmission, memory formation and synaptic plasticity. Magnetic resonance spectroscopy (MRS) studies on bipolar disorder show a number of alterations in cerebral level of GABA and glutamate in different cerebral areas when compared to healthy subjects and other mood disorders. Objective: Investigate in bipolar patients and healthy controls the association of GAD1 and Reln single nucleotide polymorphisms(SNP) and cerebral levels of GABA/glutamate on MRS. Methods: 70 symptomatic bipolar I patients medication free and 70 healthy controls are going to be genotyped for GAD1 and Reln SNPs and GABA/glutamate MRS.

Key words: GAD1, GAD67, bipolar, GABA, Glutamate, Reelin, Rln, Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder type I diagnose (DSM-IV criteria)
* Medication free (4 last weeks)

Exclusion Criteria:

* heavy smokers
* cannabis use
* recent alcohol abuse (14 days)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Bipolar Disorder Patients
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
association between GABA/glutamate brain levels and GAD1 polymorphisms | single evaluation

SECONDARY OUTCOMES:
association between GABA/glutamate brain levels and Reelin polymorphisms | single evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry HCFMUSP, São Paulo, Brazil

REFERENCES:
- [Background] Tost H, Lipska BK, Vakkalanka R, Lemaitre H, Callicott JH, Mattay VS, Kleinman JE, Marenco S, Weinberger DR. No effect of a common allelic variant in the reelin gene on intermediate phenotype measures of brain structure, brain function, and gene expression. Biol Psychiatry. 2010 Jul 1;68(1):105-7. doi: 10.1016/j.biopsych.2010.02.023. PMID 20434133
- [Background] Straub RE, Lipska BK, Egan MF, Goldberg TE, Callicott JH, Mayhew MB, Vakkalanka RK, Kolachana BS, Kleinman JE, Weinberger DR. Allelic variation in GAD1 (GAD67) is associated with schizophrenia and influences cortical function and gene expression. Mol Psychiatry. 2007 Sep;12(9):854-69. doi: 10.1038/sj.mp.4001988. Epub 2007 May 1. PMID 17767149
- [Derived] Scotti-Muzzi E, Chile T, Moreno R, Pastorello BF, da Costa Leite C, Henning A, Otaduy MCG, Vallada H, Soeiro-de-Souza MG. ACC Glu/GABA ratio is decreased in euthymic bipolar disorder I patients: possible in vivo neurometabolite explanation for mood stabilization. Eur Arch Psychiatry Clin Neurosci. 2021 Apr;271(3):537-547. doi: 10.1007/s00406-020-01096-0. Epub 2020 Jan 28. PMID 31993746
- [Derived] Soeiro-de-Souza MG, Lafer B, Moreno RA, Nery FG, Chile T, Chaim K, da Costa Leite C, Machado-Vieira R, Otaduy MC, Vallada H. The CACNA1C risk allele rs1006737 is associated with age-related prefrontal cortical thinning in bipolar I disorder. Transl Psychiatry. 2017 Apr 11;7(4):e1086. doi: 10.1038/tp.2017.57. PMID 28398341
- [Derived] Soeiro-de-Souza MG, Pastorello BF, Leite Cda C, Henning A, Moreno RA, Garcia Otaduy MC. Dorsal Anterior Cingulate Lactate and Glutathione Levels in Euthymic Bipolar I Disorder: 1H-MRS Study. Int J Neuropsychopharmacol. 2016 Aug 12;19(8):pyw032. doi: 10.1093/ijnp/pyw032. Print 2016 Aug. PMID 27207914